CLINICAL TRIAL: NCT06338865
Title: Standard vs. Lower Pressure Pneumoperitoneum in Laparoscopic Gynecologic Surgery: A Randomized Controlled Trial
Brief Title: Short Title: Standard vs. Lower Pressure Pneumoperitoneum
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Matthew Siedhoff, MD MSCR, Vice Chair for Gynecology, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Study00003146
Record Dates: First submitted 2024-03-21; First posted 2024-04-01 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Laparoscopic Surgery
Keywords: laparoscopic surgery; insufflation; pneumoperitoneum; gynecologic surgery; postoperative pain; robotic surgery
MeSH Terms: conditions — Pneumoperitoneum; Pain, Postoperative | interventions — Carbon Dioxide; Bupivacaine; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and post-anesthesia care unit nurses will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 15mmHg (Conventional Laparoscopic Arm) (Active Comparator): Standard Pressure, Conventional Laparoscopic Arm
  Interventions: Other: Carbon dioxide; Drug: Bupivacaine; Drug: Oxycodone
- 12mmHg (Conventional Laparoscopic Arm) (Experimental): Lower Pressure, Conventional Laparoscopic Arm
  Interventions: Other: Carbon dioxide; Drug: Bupivacaine; Drug: Oxycodone
- 10mmHg (Conventional Laparoscopic Arm) (Experimental): Lowest Pressure, Conventional Laparoscopic Arm
  Interventions: Other: Carbon dioxide; Drug: Bupivacaine; Drug: Oxycodone
- 15mmHg (Robotic-Assisted Laparoscopic Arm) (Active Comparator): Standard Pressure, Robotic-Assisted Laparoscopic Arm
  Interventions: Other: Carbon dioxide; Drug: Bupivacaine; Drug: Oxycodone
- 12mmHg (Robotic-Assisted Laparoscopic Arm) (Experimental): Lower Pressure, Robotic-Assisted Laparoscopic Arm
  Interventions: Other: Carbon dioxide; Drug: Bupivacaine; Drug: Oxycodone
- 10mmHg (Robotic-Assisted Laparoscopic Arm) (Experimental): Lowest Pressure, Robotic-Assisted Laparoscopic Arm
  Interventions: Other: Carbon dioxide; Drug: Bupivacaine; Drug: Oxycodone

INTERVENTIONS:
Other: Carbon dioxide — Gas used for insufflation pressure
Drug: Bupivacaine — Local subcutaneous infiltration of all port sites with 0.25% bupivacaine will be performed prior to each incision. Remaining local anesthetic will be administered into the incision sites prior to the conclusion of the case (30cc total).
Drug: Oxycodone — All patients will be prescribed a total of 10 pills of oxycodone 5mg, which is the standard amount that our practice prescribes for patients after laparoscopic surgery.

SUMMARY:
This study aims to investigate the effect of varying insufflation pressures on post-operative pain and adequacy of surgical field visualization among patients undergoing laparoscopic surgery with a minimally invasive gynecologic surgeon.

DETAILED DESCRIPTION:
This will be a single-center, single-blinded randomized controlled trial evaluating the impact of lower pressure pneumoperitoneum on post-operative pain and surgical field visualization among patients undergoing laparoscopic gynecologic surgery. The investigators hypothesize that lower insufflation pressures will decrease post-operative pain in the immediate post-operative period without compromising surgical field visualization. The study will include 3 groups corresponding to varying insufflation pressures: 15mmHg (standard), 12mmHg and 10mmHg. Participants will be 1:1:1 allocated to the 15mmHg, 12mmHg or 10mmHg groups (parallel design) by block randomization.

Given inherent differences in how pneumoperitoneum is maintained during conventional versus robotic-assisted laparoscopic surgery, the investigators will be enrolling patients in two separate arms depending on their planned procedure:

1. Standard vs. Lower Pressure Pneumoperitoneum in Conventional Laparoscopic Gynecologic Surgery
2. Standard vs. Lower Pressure Pneumoperitoneum in Robotic-Assisted Laparoscopic Gynecologic Surgery.

The methodology for the two arms will be otherwise identical.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* 18 years of age or older
* Undergoing laparoscopic surgery at Cedars-Sinai Medical Center with a surgeon in the Minimally Invasive Gynecologic Surgery division.

Exclusion Criteria:

* Pregnancy
* Urgent/non-scheduled surgery
* Scheduled for planned or possible concomitant non-gynecologic surgery (e.g., urologic or colorectal procedure)
* Baseline opioid use
* Allergy or intolerance to bupivacaine (or amide class of anesthetics), oxycodone, acetaminophen, or ibuprofen
* Planned post-operative admission

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Maximum documented pain score in post-anesthesia care unit (PACU) (numerical rating scale, 0-10) | Postoperatively, before discharge from PACU (postoperative day 0)
  The numerical rating scale is a pain screening tool that is routinely used to assess pain severity in the postoperative setting using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable."

SECONDARY OUTCOMES:
First reported pain score in PACU (numerical rating scale, 0-10) | Immediately upon arrival to PACU (postoperative day 0)
  The numerical rating scale is a pain screening tool that is routinely used to assess pain severity in the postoperative setting using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable."
Last reported pain score in PACU prior to discharge (numerical rating scale, 0-10) | Immediately prior to discharge from PACU (postoperative day 0)
  The numerical rating scale is a pain screening tool that is routinely used to assess pain severity in the postoperative setting using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable."
Inpatient morphine milligram equivalents | Day of surgery (postoperative day 0)
  Daily total of opioid medications administered on the day of surgery
Total number of 5mg oxycodone pills taken in the 2 weeks following discharge | Assessed at postoperative day 14
Need for insufflation pressure increase intra-operatively due to inadequate visualization | Intraoperative
Operative time | Intraoperative
Estimated blood loss | Intraoperative
Intraoperative complications | Intraoperative
Conversion to laparotomy | Intraoperative
Postoperative length of stay | Postoperatively, before discharge from PACU (postoperative day 0)
  From arrival to PACU to discharge home
Surgeon-reported adequacy of assigned insufflation pressure | Immediately following surgery
  Surgeons will rate their agreement with the following statement on a 5-point Likert scale (from strongly disagree to strongly agree): "The assigned insufflation pressure was adequate for this procedure"
Need for adjustment of insufflation pressure | Intraoperative
  In a post-op questionnaire, surgeons will indicate whether the insufflation pressure was adjusted at any point during the procedure (yes/no).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Siedhoff, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No